CLINICAL TRIAL: NCT00932919
Title: Thought Field Therapy and Cognitive Therapy for Agoraphobia - a Randomized Controlled Intervention Study Where the Efficacy of Thought Field Therapy is to be Compared to Cognitive Therapy
Brief Title: Thought Field Therapy and Cognitive Therapy for Agoraphobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SSHF-70343-AUIR-2
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Agoraphobia
Keywords: Agoraphobia; Cognitive therapy; Thought field therapy; Psychotherapy research
MeSH Terms: conditions — Agoraphobia | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Thought field therapy (Experimental): 24 randomly selected patients will be treated with 5 sessions of standard Thought field therapy.
  Interventions: Behavioral: Thought field therapy
- Cognitive therapy (Active Comparator): Treatment with Cognitive therapy, 12 sessions with manualized therapy according to David Clark's model.
  Interventions: Behavioral: Cognitive therapy
- Wait list (Other): 24 patients will be randomly selected to 3 months on a wait list, thereafter randomly selected to either Cognitive therapy or Thought field therapy.
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: Thought field therapy — 5 sessions with Thought field therapy
  Other Names: TFT
  Arms: Thought field therapy
Behavioral: Cognitive therapy — 12 sessions of Cognitive therapy
  Other Names: CBT
  Arms: Cognitive therapy
Behavioral: Wait list — 3 months waiting, then randomized to either thought field therapy or cognitive therapy
  Other Names: WL
  Arms: Wait list

SUMMARY:
The purpose for this study is to find out if Thought field therapy has the same effect as, or better effect than, Cognitive therapy for Agoraphobia.

DETAILED DESCRIPTION:
Thought field therapy is an alternative treatment method that has shown, by casuistic reports, to give good results when applied for anxiety disorders. In this study 72 patients will be randomized to three groups. 24 patients will receive cognitive therapy as a control method, 24 patients will receive thought field therapy. The remaining 24 patients will wait three months, and then be randomized to either of the two therapies.

Before inclusion all patients will be diagnosed with M.I.N.I. and SCID II. They will fill out self evaluation forms for symptoms and quality of life, before and after treatment, and one year after treatment.

All patients will undergo an interview with ADIS on panic and agoraphobic diagnosis and symptoms before starting treatment, and on panic and agoraphobic symptoms immediately after and one year after treatment. These interviews will be done by psychologists who are blinded for which type of treatment the patients have got.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 years or older,
* Patients with agoraphobia,
* Patients with a score on Mobility Inventory "Alone" of 2.5 or more,
* Patients who give a written consent to participate.

Exclusion Criteria:

* Psychosis (past or present),
* Drug abuse or dependency,
* Moderate or high score on suicidal behaviour on the M.I.N.I.,
* Patients who have another illness (other than panic disorder or agoraphobia) and are in need of immediate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in agoraphobic situation scores in ADIS. | Immedeately and 12 months after treatment

SECONDARY OUTCOMES:
Interference score in ADIS | Immediately and 12 months after treatment
Mobility Inventory | Immediately and 12 months after treatment
Agoraphobic Cognitions Questionnaire | Immediately and 12 months after treatment
Body Sensations Questionnaire | Immediately and 12 months after treatment
BDI | Immediately and 12 months after treatment
BAI | Immediately and 12 months after treatment
WHOQOL-BREF | Immediately and 12 months after treatment
SF-36 | Immediately and 12 months after treatment
Safety Seeking Behaviours Questionnaire. | Immediately and 12 months after treatment
Panic scale | Immediately and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Audun C Irgens, MD, Principal Investigator — Sorlandet Hospital HF, Norway
Locations (1):
- Sorlandet Hospital, Arendal, Norway

REFERENCES:
- [Derived] Irgens AC, Hoffart A, Nysaeter TE, Haaland VO, Borge FM, Pripp AH, Martinsen EW, Dammen T. Thought Field Therapy Compared to Cognitive Behavioral Therapy and Wait-List for Agoraphobia: A Randomized, Controlled Study with a 12-Month Follow-up. Front Psychol. 2017 Jun 20;8:1027. doi: 10.3389/fpsyg.2017.01027. eCollection 2017. PMID 28676782